CLINICAL TRIAL: NCT02549560
Title: Effects of the Transcranial Direct Current Stimulation on Prevention of Cognitive Dysfunction in Elderly Patients Submitted to Cardiac Surgeries: Prospective, Randomized and Double-blind Study
Brief Title: Effects of the Transcranial Stimulation on Prevention of Cognitive Dysfunction in Cardiac Surgery
Acronym: tDCS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Harvard Medical School (HMS and HSDM) (Other)
Responsible Party: Principal Investigator, Livia Stocco Sanches Valentin, Ph.D., University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Transcranial Stimulation
Record Dates: First submitted 2015-09-05; First posted 2015-09-15 (Estimated); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Postoperative Cognitive Dysfunction
Keywords: tDCS; Cardiac Surgery
MeSH Terms: conditions — Postoperative Cognitive Complications | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tDCS GROUP (Active Comparator): These patients will be submitted to 2 daily sessions of cerebral stimulation, starting from the first day after the surgery, for 4 consecutive days, with each session having 20 minutes, and a minimum break of 8 hours between them. Will be applied a direct current stimulus of 2 milliampere (mA) in the right anode and in the left cathode on the prefrontal right region.
  Interventions: Device: tDCS
- CONTROL GROUP (Sham Comparator): In these patients will be applied, with the same equipment used in tDCS, a simulated stimulus similar to the active one. They will also be submitted to some psychological test to evaluate theirs mnemonics, attentional, executive and global functions.
  Interventions: Device: tDCS

INTERVENTIONS:
Device: tDCS — Application of two daily sessions of cerebral stimulation starting from the first day after de surgery, for 4 consecutive days, with each session having 20 minutes, having an 8 hour minimum break between them. Will be applied a direct current stimulus of 2 milliampere (mA) (right anode/left cathode) in the prefrontal right region.
  Other Names: transcranial Direct Current Stimulation

SUMMARY:
Postoperative cognitive dysfunction (POCD) is a contrary event observed between 20 to 83%, especially on elderly and patients submitted to cardiac surgery. The prevention and rehabilitation on cases of POCD can improve the quality of life and decrease the mortality in surgical patients. The effect of the noninvasive cerebral stimulation, also known as transcranial Direct Current Stimulation (tDCS) has been studied to be used in the treatment of brain injuries and depression, and also in the cognitive rehabilitation. The hypothesis is that the use of the tDCS technique can decrease the occurrence of POCD and cognitively rehabilitate patients submitted to cardiac surgeries.

DETAILED DESCRIPTION:
SUMMARY Postoperative cognitive dysfunction (POCD) is a contrary event observed between 20 to 83%, especially on elderly, patients submitted to cardiac surgery. Besides the difficult diagnosis, the limitations of prevention and rehabilitation on cases of POCD may compromise the quality of life and increase the mortality in surgical patients. The neuromodulator effect of the noninvasive cerebral stimulation, also known as transcranial stimulation, with a low intensity electric current (tDCS) has been studied to be used in the treatment of brain injuries and depression, and also in the cognitive rehabilitation. The hypothesis is that the use of the tDCS technique in sessions can decrease the occurrence of POCD and cognitively rehabilitate patients submitted to cardiac surgeries. The objective of this study is to evaluate the effect of the tDCS over the occurrence of POCD on patient submitted to cardiac surgeries with cardiopulmonary bypass (CPB)

After the approval by the constitutional ethics commission, will be included in the study 138 adult patients submitted to a cardiac surgery. After the subscription of the consent form by the responsible the patients will be randomly allocated in two groups:

tDCS GROUP: These patients will be submitted to 2 daily sessions of cerebral stimulation, starting from the first day after the surgery, for 4 consecutive days, with each session having 20 minutes, and a minimum break of 8 hours between them. Will be applied a direct current stimulus of 2 milliampere (mA) in the right anode and in the left cathode on the prefrontal right region.

CONTROL GROUP: In these patients will be applied, with the same equipment used in tDCS, a simulated stimulus similar to the active one. They will also be submitted to some psychological test to evaluate theirs mnemonics, attentional, executive and global functions. The volunteers will be evaluated in a model with the intention to treat (ITT) of recovering the cognitive functions evaluated by scores on the test based on normative tables, this is the primary outcome. The secondary outcome will be improvements on the response of these cognitive tests, the admission of these patients will last 15 days in the intensive treatment unity and in the hospital. There will also be evaluated data relative to the surgery, the cognitive evolution and the quality of life in postoperative period.

Will also be applied neuropsychological tests to evaluate memory, attention, and executive functions as well as another tests to assess specifics contents useful to describe the sample and research' results.

The tests applied will be on specific data set. Sociodemographic data will be analyzed including education, marital status, occupation, and current medication. Signs and symptoms of depression will be assess preoperatively using the Beck Depression Inventory (BDI), for screening on global cognitive will be use Telephone Interview for Cognitive Status (TICS), will be use the Verbal Learning Test (VLT) for long-term memory and the Recognition Memory Test (TEM-R) for visual memory, the Symbol Digit Modified Test (SDMT) will be use to assess short-term memory, visual search skill and attention, STROOP Test will be assess the selective attention, inhibitory ability and mental flexibility that are constructs of executive function and the Trail Making Test (TMT) for the assessment of selective and alternating attention.

Beck Depression Inventory (BDI), which consists of 21 questions that explore depressive symptoms on a scale of 0 to 4, where zero represents no symptoms and four is the maximum symptomatology. A total of 14 points will be consider indicative of the presence of moderate depressive symptoms.

Patient Questionnaire health (PHQ-9), this questionnaire about the health of the patient is an instrument with 9 questions. Each question has 4 possible responses: 0 (no day), 1 (several days), 2 (more than half days), and 3 (nearly every day). The PHQ-9 can be interpreted in three ways: 10 in the form of algorithm, identifying individuals with a major depressive episode and tracking probable cases of major depressive disorder; 20 as a continuous measure, with scores between 0 and 27 points, being able to assess levels of depressive symptoms through the cut- points 5, 10, 15 and 20 points = mild depression, moderate, severe and serious; 30 as continuous measurements with scores between 0 and 27 points, classifying the individuals dichotomous through the use of a single cutting point (typically ≥10).

The Confusion Assessment Method (CAM-ICU) is a test to evaluate delirium; patients are evaluating qualitatively by the researcher from a number of simple questions to the presence or absence of postoperative delirium. This review will be done on the patient to wake up from anesthesia in the first hours after surgery and on the third day postoperative.

The Telephone Interview for Cognitive Status (TICS) will be use as a standardized test to assess neuropsychological functioning when assessing cognitive skills. This test can be used when screening personally is impractical or when patients are unable to attend the clinic. This test consists of a structured interview with 11 items that assess the skills of spatial and temporal orientation, mental control, memory, general information, language and calculations.

Memory will be assessed using the Verbal Learning Test (VLT) this test consists of a list of words. A list of 15 words is presented and must to be stored and recalled in three successive attempts (VLT / A-B-C), with delayed recall after 25 minutes (VLT-Delay). Rate is the number of words recalled and the number of errors for each presentation. The VLT evaluates the modalities of memory immediate, consolidated and long-term. This instrument will be held in two stages: pre-operative at the time of 1st evaluation before surgery and postoperatively in the second and final assessment between day 10 and 15 postoperatively.

The Recognition Memory Test (TEM-R) consists of storing pictures and words to further identify remembered stimuli. For the stimulus responses can be presented to the subject in graphic form (figures) or written (words). This instrument will be held in two stages: pre-operative at the time of 1st evaluation before surgery and postoperatively in the second and final assessment between day 10 and 15 postoperatively.

The Symbol Digit Modified Test (SDMT) will be applied for the evaluation of short-term memory, visual search skill and attention. This is a graphical task where the individual has to fill in symbols exemplified in the spaces below the corresponding number within 180 seconds. The result is measured as the number of symbols drawn and the number of errors.

Attention will be assessed by STROOP Test, which consists in presenting three paper sheets to the subject. The first one, the patient should verbalize the names of colors printed in black ink. In the second, verbalization is made of color are filled rectangles, the same provision of the words of the previous slide. The third blade consist in verbalize colors printed over the written word. Evaluates selective attention, inhibitory ability and mental flexibility that are constructs of executive function. Scores obtained include the number of words (Word task), number of bar colors (Color), and number of color words (Color-Word) completed within a set time, or as noted above, the amount of time required to complete each of the tasks. We will consider the number of errors as well.

Attention will also be evaluated using the Trail Making Test (TMT) for the assessment of selective and alternating attention. In part A of the test, the subject must draw lines connecting consecutively numbered circles. In part B, the subject must draw lines connecting circles alternately with letters and numbers in a sequence. The result is measured as time and trail errors. The Attention function will be examined with Trail Making Test (TMT). This test consists of two parts. In Part A, the subject must draw lines connecting consecutively numbered circles. In Part B, the subject must draw lines alternately connecting circles with letters and numbers in a sequence. The test involves addition of alternate and selective attention, visual screening and complex manual dexterity (Part A) and executive processes (Part B). Among the executive procedures, the inhibitory ability and cognitive alternating seem to be those most required in completing the task. They are valued the time spent and the number of errors in each of. These instrument will be held in two stages: pre-operative at the time of 1st evaluation before surgery and postoperatively in the second and final assessment between day 10 and 15 postoperatively.

The neuropsychological test will be describes according to the groups and the moments of application, with average usage, standard deviation and compared to results of normative charts with Z-score (±1,96) being the reference of cognitive dysfunction. The data will be expressed in means, medians, confidence intervals (CI-95%) and standard deviation (SD) and evaluated as to normality, being the normal data analyzed by Generalized Estimating Equation (GEE), to comparison of the results between the two groups. P<0,05 will be considered significant.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients over 18 years candidates do cardiac surgeries with extracorporeal circulation. Patients that signed the Free and Clarified Consent Form

Exclusion Criteria:

* Historic of progressive mental disease or dementia
* Psychiatric disease that affects cognition
* Lack of fluency of the Portuguese language
* Historic of epilepsies, convulsions, fainting and syncope
* With serious cranial traumas, carriers of ventriculoperitoneal derivation valves or metallic objects implanted in the brain
* With hearing problems or cochlear implants
* With cardiac pacemaker or any metallic implants in the body; Use of neuropsychiatric medications on the preoperative period
* Already submitted to the stimulation of the tDCS

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2021-07-08 (Actual); Primary Completion 2022-12-29 (Actual); Study Completion 2023-11-08 (Actual)

PRIMARY OUTCOMES:
tDCS as a cognitive enhancer for patients with postoperative cognitive dysfunction after cardiac surgery | 18 months
  Evaluate if tDCS sessions decrease the occurrence of POCD in patients submitted to extracorporeal circulation on cardiac surgery. Neuropsychological testing: Changes in results from neuropsychological assessment pre (before the first stimulation) to post treatment (after the last stimulation). There will be a eight days time frame from pre assessment to post assessment. The improvement of the skills and cognitive functions will be compare with results of tests for evaluation of quality of life, depressive symptoms and neuropsychological battery to assess, attention, visuospatial perception, immediate memory, operational, long-term memory and executive skills and recall, including processing speed.

SECONDARY OUTCOMES:
Changes in results from neuropsychological assessment pre (before the first stimulation) to post treatment (after the last stimulation). | 15 days
  Evaluate if tDCS sessions rehabilitate the compromised cognitive functions on patients submitted to extracorporeal circulation cardiac surgery. Neuropsychological testing: Changes in results from neuropsychological assessment pre (before the first stimulation) to post treatment (after the last stimulation). The improvement of the skills and cognitive functions will be compare with results of tests for evaluation of quality of life, depressive symptoms and neuropsychological battery to assess, attention, visuospatial perception, immediate memory, operational, long-term memory and executive skills and recall, including processing speed.

CONTACTS AND LOCATIONS:
Overall Officials: Livia S Valentin, Ph.D., Principal Investigator — University of Sao Paulo School of Medicine
Locations (1):
- Livia Stocco Sanches Valentin, São Paulo, Brazil

REFERENCES:
- [Background] Beck AT SR. Beck depression Inventory. manual. San Antonio: Psychology Corporation. 1993
- [Result] Nie H, Zhao B, Zhang YQ, Jiang YH, Yang YX. Pain and cognitive dysfunction are the risk factors of delirium in elderly hip fracture Chinese patients. Arch Gerontol Geriatr. 2012 Mar-Apr;54(2):e172-4. doi: 10.1016/j.archger.2011.09.012. Epub 2011 Oct 19. PMID 22014763
- [Result] van Harten AE, Scheeren TW, Absalom AR. A review of postoperative cognitive dysfunction and neuroinflammation associated with cardiac surgery and anaesthesia. Anaesthesia. 2012 Mar;67(3):280-93. doi: 10.1111/j.1365-2044.2011.07008.x. PMID 22321085
- [Result] Moller JT, Cluitmans P, Rasmussen LS, Houx P, Rasmussen H, Canet J, Rabbitt P, Jolles J, Larsen K, Hanning CD, Langeron O, Johnson T, Lauven PM, Kristensen PA, Biedler A, van Beem H, Fraidakis O, Silverstein JH, Beneken JE, Gravenstein JS. Long-term postoperative cognitive dysfunction in the elderly ISPOCD1 study. ISPOCD investigators. International Study of Post-Operative Cognitive Dysfunction. Lancet. 1998 Mar 21;351(9106):857-61. doi: 10.1016/s0140-6736(97)07382-0. PMID 9525362
- [Result] Koster S, Hensens AG, van der Palen J. The long-term cognitive and functional outcomes of postoperative delirium after cardiac surgery. Ann Thorac Surg. 2009 May;87(5):1469-74. doi: 10.1016/j.athoracsur.2009.02.080. PMID 19379886
- [Result] Martin JF, Melo RO, Sousa LP. Postoperative cognitive dysfunction after cardiac surgery. Rev Bras Cir Cardiovasc. 2008 Apr-Jun;23(2):245-55. doi: 10.1590/s0102-76382008000200015. English, Portuguese. PMID 18820789
- [Result] Monk TG, Weldon BC, Garvan CW, Dede DE, van der Aa MT, Heilman KM, Gravenstein JS. Predictors of cognitive dysfunction after major noncardiac surgery. Anesthesiology. 2008 Jan;108(1):18-30. doi: 10.1097/01.anes.0000296071.19434.1e. PMID 18156878
- [Result] Mracek J, Holeckova I, Chytra I, Mork J, Stepanek D, Vesela P. The impact of general versus local anesthesia on early subclinical cognitive function following carotid endarterectomy evaluated using P3 event-related potentials. Acta Neurochir (Wien). 2012 Mar;154(3):433-8. doi: 10.1007/s00701-011-1270-4. Epub 2012 Jan 15. PMID 22245975
- [Result] Lefrere JJ, Fine JM, Lambin P, Muller JY, Courouce AM, Salmon C. Monoclonal gammopathies in asymptomatic HIV-seropositive patients. Clin Chem. 1987 Sep;33(9):1697-8. No abstract available. PMID 3621592
- [Result] Fan Q, Cai Y, Chen K, Li W. Prognostic study of sevoflurane-based general anesthesia on cognitive function in children. J Anesth. 2013 Aug;27(4):493-9. doi: 10.1007/s00540-013-1566-z. Epub 2013 Feb 6. PMID 23386252
- [Result] Funder KS, Steinmetz J. Post-operative cognitive dysfunction - Lessons from the ISPOCD studies. Trends in Anaesthesia and Critical Care. 2012;2(3):94-7
- [Result] Laalou FZ, Jochum D, Pain L. [Postoperative cognitive dysfunction (POCD): strategy of prevention, assessment and management]. Ann Fr Anesth Reanim. 2011 Oct;30(10):e49-53. doi: 10.1016/j.annfar.2011.08.009. Epub 2011 Sep 25. French. PMID 21945705
- [Result] Newfield P. Postoperative cognitive dysfunction. F1000 Med Rep. 2009 Feb 24;1:14. doi: 10.3410/M1-14. PMID 20948768
- [Result] Crosby G, Culley DJ, Hyman BT. Preoperative cognitive assessment of the elderly surgical patient: a call for action. Anesthesiology. 2011 Jun;114(6):1265-8. doi: 10.1097/ALN.0b013e31821b1bc8. No abstract available. PMID 21490501
- [Result] DeCrane SK, Sands LP, Young KM, DePalma G, Leung JM. Impact of missing data on analysis of postoperative cognitive decline (POCD). Appl Nurs Res. 2013 May;26(2):71-5. doi: 10.1016/j.apnr.2012.11.001. Epub 2013 Jan 3. PMID 23290047
- [Result] Fletcher JM. Dyslexia: The evolution of a scientific concept. J Int Neuropsychol Soc. 2009 Jul;15(4):501-8. doi: 10.1017/S1355617709090900. PMID 19573267
- [Result] Brambati SM, Termine C, Ruffino M, Danna M, Lanzi G, Stella G, Cappa SF, Perani D. Neuropsychological deficits and neural dysfunction in familial dyslexia. Brain Res. 2006 Oct 3;1113(1):174-85. doi: 10.1016/j.brainres.2006.06.099. Epub 2006 Aug 23. PMID 16934234
- [Result] Gonzalez-Gadea ML, Baez S, Torralva T, Castellanos FX, Rattazzi A, Bein V, Rogg K, Manes F, Ibanez A. Cognitive variability in adults with ADHD and AS: disentangling the roles of executive functions and social cognition. Res Dev Disabil. 2013 Feb;34(2):817-30. doi: 10.1016/j.ridd.2012.11.009. Epub 2012 Dec 7. PMID 23220737
- [Result] Ames CS, White SJ. Are ADHD traits dissociable from the autistic profile? Links between cognition and behaviour. J Autism Dev Disord. 2011 Mar;41(3):357-63. doi: 10.1007/s10803-010-1049-0. PMID 20585847
- [Result] Gualtieri CT, Johnson LG. Medications do not necessarily normalize cognition in ADHD patients. J Atten Disord. 2008 Jan;11(4):459-69. doi: 10.1177/1087054707305314. Epub 2007 Oct 12. PMID 17934180
- [Result] Brunoni AR, Nitsche MA, Bolognini N, Bikson M, Wagner T, Merabet L, Edwards DJ, Valero-Cabre A, Rotenberg A, Pascual-Leone A, Ferrucci R, Priori A, Boggio PS, Fregni F. Clinical research with transcranial direct current stimulation (tDCS): challenges and future directions. Brain Stimul. 2012 Jul;5(3):175-195. doi: 10.1016/j.brs.2011.03.002. Epub 2011 Apr 1. PMID 22037126
- [Result] Tadini L, El-Nazer R, Brunoni AR, Williams J, Carvas M, Boggio P, Priori A, Pascual-Leone A, Fregni F. Cognitive, mood, and electroencephalographic effects of noninvasive cortical stimulation with weak electrical currents. J ECT. 2011 Jun;27(2):134-40. doi: 10.1097/YCT.0b013e3181e631a8. PMID 20938352
- [Result] Hasan A, Nitsche MA, Herrmann M, Schneider-Axmann T, Marshall L, Gruber O, Falkai P, Wobrock T. Impaired long-term depression in schizophrenia: a cathodal tDCS pilot study. Brain Stimul. 2012 Oct;5(4):475-83. doi: 10.1016/j.brs.2011.08.004. Epub 2011 Sep 5. PMID 21945231
- [Result] Zanao TA, Moffa AH, Shiozawa P, Lotufo PA, Bensenor IM, Brunoni AR. Impact of two or less missing treatment sessions on tDCS clinical efficacy: results from a factorial, randomized, controlled trial in major depression. Neuromodulation. 2014 Dec;17(8):737-42; discussion 742. doi: 10.1111/ner.12167. Epub 2014 Apr 11. PMID 24725075
- [Result] Santos MD, Gagliardi RJ, Mac-Kay AP, Boggio PS, Lianza R, Fregni F. Transcranial direct-current stimulation induced in stroke patients with aphasia: a prospective experimental cohort study. Sao Paulo Med J. 2013;131(6):422-6. doi: 10.1590/1516-3180.2013.1316595. PMID 24346782
- [Result] Fleck MP, Louzada S, Xavier M, Chachamovich E, Vieira G, Santos L, Pinzon V. [Application of the Portuguese version of the abbreviated instrument of quality life WHOQOL-bref]. Rev Saude Publica. 2000 Apr;34(2):178-83. doi: 10.1590/s0034-89102000000200012. Portuguese. PMID 10881154
- [Result] BECK AT, WARD CH, MENDELSON M, MOCK J, ERBAUGH J. An inventory for measuring depression. Arch Gen Psychiatry. 1961 Jun;4:561-71. doi: 10.1001/archpsyc.1961.01710120031004. No abstract available. PMID 13688369
- [Result] Klugkist M, Sedemund-Adib B, Schmidtke C, Schmucker P, Sievers HH, Huppe M. [Confusion Assessment Method for the Intensive Care Unit (CAM-ICU): diagnosis of postoperative delirium in cardiac surgery]. Anaesthesist. 2008 May;57(5):464-74. doi: 10.1007/s00101-008-1356-4. German. PMID 18345523
- [Result] Baccaro A, Segre A, Wang YP, Brunoni AR, Santos IS, Lotufo PA, Bensenor IM, Goulart AC. Validation of the Brazilian-Portuguese version of the Modified Telephone Interview for cognitive status among stroke patients. Geriatr Gerontol Int. 2015 Sep;15(9):1118-26. doi: 10.1111/ggi.12409. Epub 2014 Nov 19. PMID 25407304
- [Result] Cavaco S, Goncalves A, Pinto C, Almeida E, Gomes F, Moreira I, Fernandes J, Teixeira-Pinto A. Auditory Verbal Learning Test in a Large Nonclinical Portuguese Population. Appl Neuropsychol Adult. 2015;22(5):321-31. doi: 10.1080/23279095.2014.927767. Epub 2015 Jan 12. PMID 25580839
- [Result] Tombaugh TN. Trail Making Test A and B: normative data stratified by age and education. Arch Clin Neuropsychol. 2004 Mar;19(2):203-14. doi: 10.1016/S0887-6177(03)00039-8. PMID 15010086